CLINICAL TRIAL: NCT02564289
Title: Cardiovascular Effects of Chronic Snus Use
Acronym: CHROS
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Jenny Bosson, MD, PhD, Umeå University
Other Study IDs: 2015/70-31
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Vascular Complications; Vascular Stiffness; Tobacco Dependence
Keywords: microvesicles, microparticles; Plethysmography; Snus; Arterial Stiffness; EPC
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples, Urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Chronic snus users: Healthy subjects that used snus for more than 15 years.
- Healthy Controls: Healthy subjects that are never-users of snus.

SUMMARY:
The current study proposes to investigate the effects of chronic snus use on the blood vessels. Several cardiovascular endpoints are measured using various methods in healthy daily snus users as well as in healthy matched controls.

DETAILED DESCRIPTION:
The Swedish moist oral snuff known as "snus" has previously been found primarily in Scandinavia. In Sweden approximately 1 in 5 men are habitual users of snus. It is estimated that 3-4% of the female population are regular users. However, the last few years has seen a shift in the global tobacco industry towards finding novel ways of entering the smokeless tobacco (ST) markets. In the United States both Camel and Marlboro brands, among others, have launched an array of ST products similar to Swedish snus. Since its launch in 2007, the US snus market has continued to grow at an exponential rate and now sells approximately 50 million cans a year.

Smoking has been studied extensively and been undoubtedly linked to a range of detrimental health effects, including cardiovascular disease. As snus has until recently been available in a limited Scandinavian market, few experimental and epidemiological studies have been performed.

A recent meta-analysis found snus to be associated with heart failure and higher risk of fatal myocardial infarctions and stroke. Following myocardial infarction, discontinuation of snus use was associated with a 50% decreased risk of mortality.

With new emerging markets worldwide publicizing the product as a discrete and healthier alternative to cigarettes, it has become all the more imperative to study the health effects of this smokeless tobacco. Using well validated methods the investigators intend to study the possible effects of chronic snus use on vascular endothelial function, thrombosis, circulating microparticles in blood and arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Normal clinical examination
* Normal ECG
* Normal routine blood test including serum lipids and HbA1C

Exclusion Criteria:

* Any form of cardiovascular disease
* Any form of systemic or chronic disorder like rheumatologic or metabolic diseases.
* Active allergy within 4 weeks of the study
* Symptoms of infection or inflammation within 4 weeks of the study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 healthy non-smoking males with regular snus consumption and 25 healthy non-smoking and non-snus using. Healthy volunteers were recruited in Umeå and surrounding communities.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Venous occlusion plethysmography | 1 day
  Venous occlusion plethysmography is a semi-invasive method of estimating vascular function in which brachial forearm blood flow is measured. In combination with intra-arterial infusion of substances with vasodilatory effects (for example bradykinin, sodium nitroprusside and acetylcholine) this method is considered the "golden standard" for assessing endothelial function. Measurements are given in ml/100 ml tissue/min.

SECONDARY OUTCOMES:
Circulating microvesicles | 1 day
  Blood sample, expressed in 10^6MVs/L
Endothelial progenitor cells | 1 day
  Blood sample, measured as CD34+KDR+(KDR:vascular endothelial growth factor receptor 2) double positive cells, and results are presented as the number of EPC events.
Arterial Stiffness | 1 day
  PWA, PWV. Expressed as Pulse wave velocity (m/s) och augmentation index adjusted for pulse 75 (%).

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Bosson, MD,PhD, Principal Investigator — Umeå University
Locations (1):
- Dept of Medicine, Lung and Allergy section, University Hospital, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hergens MP, Alfredsson L, Bolinder G, Lambe M, Pershagen G, Ye W. Long-term use of Swedish moist snuff and the risk of myocardial infarction amongst men. J Intern Med. 2007 Sep;262(3):351-9. doi: 10.1111/j.1365-2796.2007.01816.x. PMID 17697156
- [Background] Bolinder G, Alfredsson L, Englund A, de Faire U. Smokeless tobacco use and increased cardiovascular mortality among Swedish construction workers. Am J Public Health. 1994 Mar;84(3):399-404. doi: 10.2105/ajph.84.3.399. PMID 8129055
- [Background] Rohani M, Agewall S. Oral snuff impairs endothelial function in healthy snuff users. J Intern Med. 2004 Mar;255(3):379-83. doi: 10.1046/j.1365-2796.2003.01279.x. PMID 14871462
- [Background] Boffetta P, Straif K. Use of smokeless tobacco and risk of myocardial infarction and stroke: systematic review with meta-analysis. BMJ. 2009 Aug 18;339:b3060. doi: 10.1136/bmj.b3060. PMID 19690343
- [Background] Arefalk G, Hambraeus K, Lind L, Michaelsson K, Lindahl B, Sundstrom J. Discontinuation of smokeless tobacco and mortality risk after myocardial infarction. Circulation. 2014 Jul 22;130(4):325-32. doi: 10.1161/CIRCULATIONAHA.113.007252. Epub 2014 Jun 23. PMID 24958793
- [Background] Arefalk G, Hergens MP, Ingelsson E, Arnlov J, Michaelsson K, Lind L, Ye W, Nyren O, Lambe M, Sundstrom J. Smokeless tobacco (snus) and risk of heart failure: results from two Swedish cohorts. Eur J Prev Cardiol. 2012 Oct;19(5):1120-7. doi: 10.1177/1741826711420003. Epub 2011 Aug 9. PMID 21828223
- [Background] Mobarrez F, Antoniewicz L, Bosson JA, Kuhl J, Pisetsky DS, Lundback M. The effects of smoking on levels of endothelial progenitor cells and microparticles in the blood of healthy volunteers. PLoS One. 2014 Feb 28;9(2):e90314. doi: 10.1371/journal.pone.0090314. eCollection 2014. PMID 24587320